CLINICAL TRIAL: NCT03527368
Title: The Time-Restricted Intake of Meals Study: A Randomized, Controlled Feeding Study
Brief Title: The Time-Restricted Intake of Meals Study
Acronym: TRIM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: American Heart Association (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IRB00155640; 17SFRN33590069 (Other Grant/Funding Number: American Heart Association)
Record Dates: First submitted 2018-05-04; First posted 2018-05-17 (Actual); Last update posted 2021-05-17 (Actual); Status verified 2021-05

CONDITIONS: PreDiabetes; Obesity
MeSH Terms: conditions — Prediabetic State; Obesity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Time-restricted feeding (Experimental)
  Interventions: Behavioral: Time-restricted feeding
- Usual feeding pattern (Other): Comparison
  Interventions: Behavioral: Usual feeding pattern

INTERVENTIONS:
Behavioral: Time-restricted feeding — Participants consume food earlier in the day
  Arms: Time-restricted feeding
Behavioral: Usual feeding pattern — Participants consume food later in the day
  Arms: Usual feeding pattern

SUMMARY:
TRIM is a randomized, controlled feeding study to evaluate if eating earlier in the day vs. later in the day impacts weight and glucose homeostasis.

ELIGIBILITY:
Inclusion Criteria:

* Prediabetes defined by HbA1c 5.7-6.4%, or type 2 diabetes with HbA1c 6.5-6.9%
* Class I-III obesity (BMI 30-50 kg/m2)
* If on medications for hypertension, stable regimen for at least past 6 months
* Willingness to adjust timing of feeding
* Willingness and ability to eat study diet and nothing else during run-in and intervention
* Willingness to complete measurement procedures

Exclusion Criteria:

* Moderate to severe obstructive sleep apnea
* Shift work;
* Other sleep/circadian disorders: e.g., circadian phase delay or phase advance; restless legs syndrome, insomnia, narcolepsy, habitual sleep <6 hours/night
* Routinely ate within compressed time window in the past year (e.g., routinely eats all food within an 10-hour or narrower window, follows an intermittent fasting protocol)
* Renal dysfunction (estimated Glomerular Filtration Rate (GFR) <30 using the simplified Chronic Kidney Disease (CKD) Epidemiology Collaboration (EPI) equation 34)
* Use of glucose-lowering medications, weight loss medications, medications for sleep disorders (sedative/hypnotic drugs, stimulants), lithium, systemic corticosteroids, diuretics, blood thinners requiring regular monitoring (e.g. warfarin), anti-psychotic drugs and antiretroviral therapy
* Body weight >400 pounds (limitation of facility scales)
* >1 drink per day of alcohol
* Active substance use disorder or significant psychiatric/psychologic disorder that would interfere with participation
* Significant food allergies, preferences, intolerances, or dietary supplements that would interfere with diet adherence
* Weight loss or gain of ≥5% during past 6 months
* Pregnant, planning to become pregnant, or breastfeeding
* Planning to start a weight loss program
* Planning to leave the area prior to end of study
* Current participation in another clinical trial
* Cancer diagnosis requiring active treatment in past two years or planned treatment (with exception of localized non-melanoma skin cancer)
* Active inflammatory bowel disease, malabsorption, or history of major gastrointestinal surgery involving bowel resection
* Myocardial infarction or stroke in past 6 months
* Prior bariatric surgery
* Any serious illness that would interfere with participation
* Other conditions or situations at the discretion of the PI

Ages: 21 Years to 69 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2018-09-24 (Actual); Primary Completion 2019-12-23 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Weight Change | 12 weeks
  Weight change will be measured in kg

SECONDARY OUTCOMES:
Fasting glucose | 12 weeks
  Change in fasting glucose
HOMA-IR | 12 weeks
  Change in HOMA-IR
AUC glucose | 12 weeks
  Area-under-the-curve for glucose on OGTT
Glycated albumin | 12 weeks
  Glycated albumin

CONTACTS AND LOCATIONS:
Overall Officials: Nisa Maruthur, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins ProHealth, Baltimore, Maryland, United States

REFERENCES:
- [Derived] Duan D, Pham LV, Jun JC, Turkson-Ocran RA, Pilla SJ, Clark JM, Maruthur NM. Effects of time-restricted eating on actigraphy-derived sleep parameters: post hoc analysis of a randomized, isocaloric feeding study. Sleep. 2025 Sep 9;48(9):zsaf089. doi: 10.1093/sleep/zsaf089. PMID 40241264
- [Derived] Maruthur NM, Pilla SJ, White K, Wu B, Maw MTT, Duan D, Turkson-Ocran RA, Zhao D, Charleston J, Peterson CM, Dougherty RJ, Schrack JA, Appel LJ, Guallar E, Clark JM. Effect of Isocaloric, Time-Restricted Eating on Body Weight in Adults With Obesity : A Randomized Controlled Trial. Ann Intern Med. 2024 May;177(5):549-558. doi: 10.7326/M23-3132. Epub 2024 Apr 19. PMID 38639542